CLINICAL TRIAL: NCT03979092
Title: Interprofessional Advanced Cardiac Life Support Training on Collaborative Skills, Self-Efficacy And Emotion Regulation: A Prospective Interventional Trial
Brief Title: Interprofessional Advanced Cardiac Life Support Training on Collaborative Skills, Self-Efficacy And Emotion Regulation
Acronym: IP-ACLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Lau Ying, Assistant Professor, National University of Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TEG AY2016/2017
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Self Efficacy; Collaborative Skills; Emotion Regulation
Keywords: Collaborative skills; Emotion regulation; Self-efficacy; Interprofessional education; Advanced Cardiac Life Support; Nursing students
MeSH Terms: conditions — Emotional Regulation | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IP-ACLS (Experimental)
  Interventions: Behavioral: IP-ACLS
- Waitlist (Other)
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: IP-ACLS — Three senior consultants and 12 trainers conduct 2-day IP-ACLS training.
  1. Pre-class activities: preparation First exposure reading on provider manual and lecturer notes about a new knowledge of ACLS to enhance self-directed learning.
  2. Interactive lecture sessions: 10 topics Interactive lectures (15-20 minutes per topic) introduce a new knowledge, which anchor to their existing knowledge according to ACLS algorithms.
  3. Simulation sessions: 10 sessions Skill sessions (50 minutes per session) used high-fidelity simulation mannequin in a team approach. Students learn through role-playing with different practical scenarios. Experiential learning is focused on hands-on and collaborative strategies for enhancing a deeper learning.
  4. Debriefing: feedback and reflection Trainers provide immediate feedback and discussion throughout the scenarios. Debriefing is focused on the positive aspect and areas for improvement.
  Arms: IP-ACLS
Behavioral: Waitlist — Waitlist group will participate in subsequent IP-ACLS training.
  Arms: Waitlist

SUMMARY:
The aim of this study is to study the effectiveness of interprofessional advanced cardiac life support (IP-ACLS) training in improving collaborative skills, self-efficacy and emotion regulation among fourth-year nursing students using a prospective, open-label, non-randomized controlled design.

The investigators hypothesized that students who participated in the IP-ACLS training are more likely to have better:

1. collaborative skills
2. self-efficacy
3. emotion regulation.

DETAILED DESCRIPTION:
A total sample size of 120 fourth year nursing students will be used. Subjective measures and objective measure are used. Principal Investigator or trained part-time undergraduate student research assistants will recruit nursing students in scheduled identical sessions. Informed consent will be obtained after an explanation of the nature, purpose, and potential risks of the study according to the information sheet.

Pre-test was conducted before starting the IP-ACLS training on Day 1; post-test 1 was conducted immediately after the IP-ACLS training on Day 2; post-test 2 was conducted 1 month after the IP-ACLS training before or after their scheduled lecture break. The students were asked to complete the self-report questionnaire in approximately 10-15 min before and after 2-day IP-ACLS workshop and 1 month follow-up.

Assessment of Interprofessional Team Collaboration Scale (AITCS), General Self-Efficacy Scale (GSE) and Emotion Regulation Questionnaire (ERQ) were used to measure collaborative skill, self-efficacy and emotion regulation using self-administration.

The Kolmogorov-Smirnov test was used to check whether the scores followed normal distributions. Independent sample t test was used for normally distributed data, whereas Mann-Whitney U test was used for non-normally distributed data to compare the AITCS, GSE and ERQ scores in two groups.

ELIGIBILITY:
Inclusion Criteria:

* National University Singapore 4th year nursing students
* Participate in the IP-ACLS training in Academic Year 2016/2017 to Academic Year 2018/2019
* Obtained informed consent

Exclusion Criteria:

* Serious psychological problems
* Cannot provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Assessment of Interprofessional Team Collaboration Scale (AITCS) | 3 years
  It consists of 37 items with 3 subscales including partnership (19 items), cooperation (11 items) and coordination (7 items) (Orchard, King, Bezzina, 2012).
  Items incorporated on a five-point Likert scale (with 5 = always, 4 = most of the time, 3 = occasionally, 2 = rarely, and 1 = never) allowing respondents to rate their current feeling about their team and themselves.
  The sum score ranged from 37 to 185. The higher the scores obtained, the more collaborative skills had.
General Self-Efficacy Scale (GSE) | 3 years
  This is a 10-item, 4-point unidimensional scale. Items had a response range from 1 (not at all true) to 4 (exactly true) (Schwarzer & Jerusalem, 1995).
  The sum scores ranged from 10 to 40. The higher the total score, the more self-efficacious the respondent.
Emotion Regulation Questionnaire (ERQ) | 3 years
  Used to measure emotion regulation which consists of two scales corresponding to two different emotion regulation strategies: cognitive reappraisal (6 items) and expressive suppression (4 items) (Gross & John, 2003).
  The 10 items are rated on a 7-point-Likert scale from strongly disagree to strongly agree. The sum score ranged from 10 to 70, participants with higher total score have better emotion regulation.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

REFERENCES:
- [Background] Orchard CA, King GA, Khalili H, Bezzina MB. Assessment of Interprofessional Team Collaboration Scale (AITCS): development and testing of the instrument. J Contin Educ Health Prof. 2012 Winter;32(1):58-67. doi: 10.1002/chp.21123. PMID 22447712
- [Background] Schwarzer R, Jerusalem M. General Self-Efficacy scale. In: Weinman J, Wright S, Johnston M, eds. Measures in health psychology: A user's portfolio. Windsor, UK: NFER-NELSON; 1995:35 - 37
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575